CLINICAL TRIAL: NCT05248737
Title: Empowering and Transforming the US Broiler Production for Growth, Profit and Sustainability
Brief Title: Bioavailability of Vitamin D(25(OH)D) and Omega-3 Fatty Acid (DHA) Enhanced Chicken
Status: Active, not recruiting | Type: Observational
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1904008786
Record Dates: First submitted 2022-02-07; First posted 2022-02-21 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Nutrition, Healthy
Keywords: Vitamin D; Omega-3 fatty acids
MeSH Terms: interventions — Eggs

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- DHA bioenhanced poultry/eggs or non-fortified poultry/eggs: In this study a group of individuals will be recruited and randomized to participate in a crossover comparing DHA enhanced poultry or control (non-fortified) poultry or to compare DHA enhanced eggs to control (non-fortified) eggs.
  Group 1: Participants will be asked to consume two meals of chicken, one meal will contain chicken that has been fed omega-3 fatty acids so the chicken contains omega 3 (DHA/EPA) fatty acids, together with a placebo, and the other meal will consist of non enhanced chicken and a DHA supplement.
  Group 2: Participants will be asked to consume two meals of eggs, one meal will contain DHA bioenhanced eggs, together with a placebo, and the other meal will consist of non enhanced eggs and a DHA supplement.
  Each participant will be asked to eat both of these forms of chicken in random order. Each study is expected to take 9-hours and the two visits will be separated by a period of two weeks. A total of 5 blood samples will be collected over a 9-h period.
  Interventions: Dietary Supplement: DHA/EPA fortified chicken plus Placebo; Dietary Supplement: non-DHA bio-enhanced chicken plus supplement DHA Omega-3; Dietary Supplement: Dietary Supplement: DHA/EPA fortified eggs plus Placebo; Dietary Supplement: non-DHA bio-enhanced eggs plus supplement DHA Omega-3
- 25(OH)D bioenhanced poultry and eggs: 25D3 Group: Weeks 0-4: Consume 5 weekly servings of 25(OH)D-enhanced chicken (300 g/serving; 1,500 g/week) + daily placebo Weeks 5-8: + additional 5 weekly 25(OH)D-enhanced eggs
  Placebo Group:
  Weeks 0-4: Consume 5 weekly servings of control chicken + daily placebo Weeks 5-8: + additional 5 weekly control eggs
  D3 Group:
  Weeks 0-4: Consume 5 weekly servings of control chicken + daily vitamin D3 (1000 IU).
  Weeks 5-8: + additional 5 weekly control eggs
  Participation in the study is expected to last 8 weeks. Individuals will be asked to come to the Human Metabolic Research Unit (HMRU) on the Cornell campus each week to pick up weekly food supplies. At five timepoints during the 8-week study, a blood draw will be collected to measure vitamin D status and other markers (e.g., hemoglobin, hematocrit, blood lipids). Each blood draw visit will take approximately 30 minutes. The total estimated time for all study visits at the HMRU is 6-7 hours over the 8-week period.
  Interventions: Dietary Supplement: non-25(OH)D fortified chicken/eggs plus vitamin D3 supplement; Dietary Supplement: 25(OH)D bioenhanced chicken and eggs plus placebo; Other: non-25(OH)D fortified chicken/eggs plus placebo

INTERVENTIONS:
Dietary Supplement: DHA/EPA fortified chicken plus Placebo — For participants who received DHA/EPA fortified chicken
  Groups: DHA bioenhanced poultry/eggs or non-fortified poultry/eggs
Dietary Supplement: non-25(OH)D fortified chicken/eggs plus vitamin D3 supplement — Provided to participants in the group where they consumed non-fortified chicken/eggs
  Groups: 25(OH)D bioenhanced poultry and eggs
Dietary Supplement: non-DHA bio-enhanced chicken plus supplement DHA Omega-3 — Used in the crossover part of the study given to the group who did not received DHA bio-enhanced chicken
  Groups: DHA bioenhanced poultry/eggs or non-fortified poultry/eggs
Dietary Supplement: 25(OH)D bioenhanced chicken and eggs plus placebo — participants will receive 25(OH)D bioenhanced chicken and eggs plus a placebo as a dietary intervention
  Groups: 25(OH)D bioenhanced poultry and eggs
Dietary Supplement: Dietary Supplement: DHA/EPA fortified eggs plus Placebo — For the participants who received DHA/EPA fortified eggs
  Groups: DHA bioenhanced poultry/eggs or non-fortified poultry/eggs
Dietary Supplement: non-DHA bio-enhanced eggs plus supplement DHA Omega-3 — for the participants who received non-DHA bio-enhanced eggs plus supplement DHA Omega-3
  Groups: DHA bioenhanced poultry/eggs or non-fortified poultry/eggs
Other: non-25(OH)D fortified chicken/eggs plus placebo — Provided to participants in the group where they consumed non-fortified chicken/eggs + placebo pills
  Groups: 25(OH)D bioenhanced poultry and eggs

SUMMARY:
The purpose of the research is to evaluate if chicken or eggs obtained from chickens that are fed a diet that contains omega-3 fatty acids (DHA/EPA), or vitamin D (as 25(OH)D) provides additional health benefits by improving the status of omega-3 fatty acids or 25(OH)D in healthy adults who eat this bioenhanced chicken or eggs.

DETAILED DESCRIPTION:
The 2015-2020 Dietary Guidelines advocate intake of lean proteins (such as chicken and fish) while limiting intake of saturated fat. Chicken contains similar protein to beef or pork but has less saturated fat. However, chicken, like other terrestrial meats, has little omega-3 polyunsaturated fatty acids such as docosahexaenoic acid (DHA) or eicosapentaenoic acid (EPA) and relatively little vitamin D. Vitamin D insufficiency is common in the US and globally, and has been linked to a number of adverse health outcomes. Vitamin D is ingested primarily from fortified dairy products, but recent animal studies have increased the D content of pork and beef, and the DHA content of chicken and of eggs produced from bioenhanced chickens. Moreover, sunlight exposure alone can enhance the 25(OH)D content of chicken. Notably, supplemental 25(OH)D is more effective than vitamin D at improving vitamin D status in humans, but little is known about the bioavailability of 25(OH)D or DHA/EPA enhanced chicken (muscle) or in enhanced eggs produced from supplemented chickens.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* Non-smoking
* Age between 18- 35 yo
* Females: premenopausal and not pregnant or lactating
* Body mass index (BMI) between 18 - 30 kg/m2.
* No preexisting medical complications (such as eating disorders, gastrointestinal disorders, malabsorption diseases, or taking medications known to influence iron homeostasis)

Exclusion Criteria:

* BMI <18 or > 30 kg/m2,
* Age <18 y or > 50y,
* Smoking
* Pregnancy, lactating
* Have gastrointestinal disorders/malabsorption diseases/dietary restrictions/medication use of medications known to impact DHA/EPA or Vitamin D 25(OH)D absorption
* Take vitamin and mineral supplementations

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults from Ithaca, NY
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2021-12-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of plasma DHA concentrations | Baseline, and time course of 1 hour, 2 hour, 4 hour and 8 hour post meal
  Measuring plasma DHA concentration across different time points to assess DHA bioavailability and absorption
Concentrations of serum 25(OH)D, vitamin D2, vitamin D3, 1,25(OH)2D and 24,25(OH)2D3 and vitamin D binding protein | Baseline, and time course of week 2, week 4, week 6, week 8
  Measuring serum 25(OH)D concentration across different time points to assess 25(OH)D bioavailability and absorption

CONTACTS AND LOCATIONS:
Locations (1):
- Human Metabolic Research Unit, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No